CLINICAL TRIAL: NCT01278758
Title: A Multi-center, Open-label, Dose-escalation Study to Assess the Pharmacokinetics of Intravenous ASA404 in Adult Advanced Cancer Patients With Impaired Renal Function and With Normal Renal Function
Brief Title: A Dose-escalation Pharmacokinetic Study of Intravenous ASA404 in Adult Advanced Cancer Patients With Impaired Renal Function and Patients With Normal Renal Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A2109; EudraCT 2009-017159-88 (Registry Identifier: EudraCT)
Record Dates: First submitted 2011-01-16; First posted 2011-01-19 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2012-11

CONDITIONS: Metastatic Cancer
Keywords: Advanced or metastatic cancer,; refractory,; core phase,; extension phase,; dose escalation,; standard chemotherapy,; doctaxel,; paclitaxel,; carboplatin,; safety,; tolerability
MeSH Terms: conditions — Neoplasm Metastasis | interventions — vadimezan

ARMS (1):
- ASA404 + standard therpy (Experimental)
  Interventions: Drug: ASA404, DMXAA or DXAA

INTERVENTIONS:
Drug: ASA404, DMXAA or DXAA

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of ASA404 in patients with refractory or relapsed metastatic cancer with impaired renal function and with normal renal function. It is very possible that patients with renal impairment will show differences in renal excretion of parent ASA404 and its metabolites, warranting a study that leads to a better pharmacokinetic assesssment in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients having histologically-proven solid tumors, who are either refractory to standard chemotherapy;
* Patients whom chemotherapy with an investigaional agent in combination with docetaxel, or paclitaxel + carboplatin is appropriate;
* Creatinine clearance according to Cockcroft-Gault formula : Normal > 80 mL/min, Mild 50-80 mL/min, Moderate 30-<50 mL/min;
* A minimum of 4 weeks must have elapsed since the last treatment with other cancer therapies;
* Potassium, calcium, magnesium and phosphorus values within the normal range;
* Body Mass Index (BMI) must be within the range of 18 and 30

Exclusion Criteria:

* Patients having CNS metastases, must have a CT or MRI of the brain performed to rule out CNS metastases;
* Patients with leptomeningeal disease metastases;
* Radiotherapy </- weeks prior to starting study drug;
* Major surgery </ 4 weeks prior to the start of study;
* Administration of CYP1A2 and CYP3A4/5 enzyme inducing or inhibiting drugs within 14 days prior to starting study drug;

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the pK of a single intravenous dose of ASA404 1200 and 1800 mg/m2 monotherapy in adult cancer patients with impaired renal function compared to matching patients with normal renal function | 12 months

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of a single i.v. dose of ASA 1200 and 1800 mg/m2 +chemotherapy (doctaxel or paclitaxel + carboplatin) in adult cancer patients with impaired renal function compared to matching patients with normal renal function | 12 months
To assess the safety and tolerability of ASA404 in adult cancer patients with impaired renal function compared to matching patients with normal renal function | 12 months
To assess the safety and tolerability of ASA404 1200 or 1800 mg/m2 in combination with chemotherapy (docetaxel or paclitaxel + carboplatin)
To evaluate ASA404 pharmacokinetic parameters including AUC (0-t last),), AUC (0-inf)), T ((½)), CL, V(Z), Cmax, and Tmax
To evaluate renal clearance (CLR) of ASA404.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Investigative Site
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Cancer Center, Hematology/Oncology Dept., Indianapolis, Indiana
  - Hematology /Oncology Associates, Rockville, Maryland
  - Joseph Ford Cancer Center/Clinical Trials Office, Henry Ford Health System, Detroit, Michigan
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- See also: Results for CASA404A2109 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5426